CLINICAL TRIAL: NCT01981252
Title: Evaluation of the Safety and Efficacy of the Ulthera® System for Wrinkle Reduction in the Peri-orbital and Peri-oral Regions
Brief Title: Peri-orbital and Peri-oral Wrinkle Reduction Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-137
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2014-10

CONDITIONS: Peri-orbital Wrinkles; Peri-oral Wrinkles
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Micro-focused Ultrasound with Visualization (MFU-V)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulthera® System Treatment (Experimental): Ulthera® System treatment of the peri-orbital and peri-oral regions.
  Interventions: Device: Ulthera® System Treatment

INTERVENTIONS:
Device: Ulthera® System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy®

SUMMARY:
This is prospective, multi-center, single-blinded, non-randomized clinical trial. Enrolled subjects will receive two Ulthera® treatments on the peri-orbital and peri-oral regions, each treatment provided 30 days apart. Follow-up visits will occur at 90 and 180 days following treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 75 years.
* Subject in good health.
* BMI<25
* Fitzpatrick wrinkle score of 3-7 in the peri-orbital and peri-oral areas.
* Moderate skin laxity in the peri-orbital area contributing to rhytids as assessed by the investigator.
* Understands and accepts the obligation not to undergo any other procedures, including neurotoxin and filler treatments, on the face through the follow-up period.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID, and Vitamin E in the 2 weeks prior to each study treatment.
* Willingness and ability to continue with their current daily skin care routine, with the exception of any use of products containing glycolic acid, for the duration of the study.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control during the study.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* BMI equal to or greater than 25
* Severe solar elastosis.
* Excessive subcutaneous fat in the area(s) to be treated.
* Mild or severe skin laxity on the area(s) to be treated.
* Significant scarring in the area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Active implantables (e.g., pacemakers or defibrillators) or metallic implants in the treatment area.
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within 4 weeks prior to study participation or during the study.
* Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* History of Bell's Palsy or epilepsy.
* History of diabetes.
* Has a known allergy, or a known history of sensitivity, to lidocaine, tetracaine, para-aminobenzoic acid (PABA).
* Concomitant therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* History of the following cosmetic treatments in the area(s) to be treated:

  1. Skin tightening procedure within the past year;
  2. Injectable fillers of any type within the past 12 or 24 months, depending on type;
  3. Neurotoxins within the past six months;
  4. Ablative resurfacing laser treatment;
  5. Nonablative, rejuvenative laser or light treatment within the past six months;
  6. Surgical dermabrasion or deep facial peels;
  7. Facelift, blepharoplasty, or browlift within the past 2 years; or
  8. Any history of contour threads.
* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Topical Retinoids within the past four weeks;
  3. Antiplatelet agents/Anticoagulants;
  4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with reduction in peri-orbital and/or peri-oral wrinkles at 90 days post-treatment #2. | Participants will be followed to 90 days post-treatment #2
  Assessment of improvement, in a blinded fashion, using the Fitzpatrick Wrinkle Scale at 90 days post-treatment #2.

SECONDARY OUTCOMES:
Number of participants with reduction in peri-orbital and/or peri-oral wrinkles at 180 days Post Treatment #2. | Participants will be followed to 180 days post-treatment #2
  Assessment of improvement, in a blinded fashion, using the Fitzpatrick Wrinkle Scale at 180 days post-treatment #2.
Number of participants with a reduction in peri-orbital and/or peri-oral wrinkle depth at 90 days post treatment #2. | Participants will be followed to 90 days post-treatment #2
  Quantitative wrinkle depth measurements will be performed using a 3-D imaging system at 90 days post-treatment #2.
Number of participants with a reduction in peri-orbital and/or peri-oral wrinkle depth at 180 days Post Treatment #2. | Participants will be followed to 180 days post-treatment #2
  Quantitative wrinkle depth measurements will be performed using a 3-D imaging system at 180 days post-treatment #2.
Overall Aesthetic Improvement | Participants will be followed to 90 days post-treatment #2
  Overall aesthetic improvement at 90 days post treatment #2 compared to baseline will be assessed using the Global Aesthetic Improvement Scale (GAIS).
Overall Aesthetic Improvement | Participants will be followed to 180 days post-treatment #2
  Overall aesthetic improvement at 180 days post treatment #2 compared to baseline will be assessed using the Global Aesthetic Improvement Scale (GAIS).
Subject Satisfaction | Participants will be followed to 90 days post-treatment #2
  Subject satisfaction will be measured at using a Patient Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Biesman, MD, Principal Investigator — Nashville Centre for Laser and Facial Surgery
Locations (5):
- United States (5):
  - Center for Advanced Facial Plastic Surgery, Beverly Hills, California
  - Aesthetic Plastic Surgical Institute, Laguna Beach, California
  - About Skin Dermatology and DermSurgery, PC, Englewood, Colorado
  - Dermatology Research Institute, Coral Gables, Florida
  - Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee